CLINICAL TRIAL: NCT05600478
Title: Physical Therapy in the Intensive Care Unit: A Comparative Study of Three Asian Countries
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other); Mariano Marcos State University (Other); Juntendo University (Other)
Responsible Party: Principal Investigator, Yu-Jung Cheng, Associate Professor, China Medical University, Taiwan
Other Study IDs: CMUH110-REC1-192
Record Dates: First submitted 2022-07-31; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: ICU
Keywords: Physiotherapy; Intensive care unit; ICU physical therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Japan: A group of ICU physical therapists working in Japan.
- Philippines: A group of ICU physical therapists working in the Philippines.
- Taiwan: A group of ICU physical therapists working in Taiwan.

SUMMARY:
This descriptive-comparative study has explored and presented an overview of the extent of PT practice in the ICU in JP, PH, and TW. Specifically, the socio-demographic and ICU-related profiles of physical therapists (PTs) in Japan (JP), Philippines (PH), and Taiwan (TW) were presented, with the inclusion of the common PT interventions and challenges encountered in delivering PT services in the ICU in the said countries.

Included in the socio-demographic variables are the respondents' sex, age, highest educational attainment, PT work experience, and hospital affiliation. As to the ICU-related variables, it includes the respondents' ICU work experience, the types of ICU where respondents primarily work, the hiring department they belong to, the status of ICU posting, the duration of ICU posting, the daily ICU stay of the respondents, their engagement in on-call ICU PT services, the usual source of ICU patient referral, the number of daily ICU patients, the ratio of PT to ICU patients, and the level of participation in ICU-related PT training. Furthermore, different interventions that are commonly implemented and challenges that are commonly encountered in ICU PT service delivery in Japan, Philippines, and Taiwan were also investigated.

DETAILED DESCRIPTION:
Physical therapy (PT) is proven beneficial among critically ill patients. However, there is an extent to the practice of PT in the intensive care unit (ICU) which differs between countries. With this, the extent of PT practice in the ICU in three Asian countries, namely Japan (JP), Philippines (PH), and Taiwan (TW), was determined and compared by specifically determining the socio-demographic and ICU-related profile of physical therapists (PTs) who have worked in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapists who:

  1. are currently residing or working in Japan, Philippines, and Taiwan;
  2. are working, or have worked in an ICU in JP, PH, or TW, and have provided PT services to critically ill patients regardless of age, sex, nationality/race, and years of work experience (in general);
  3. have an active e-mail address; and
  4. provided informed consent

Exclusion Criteria:

* Physical therapists who are:

  1. newly hired (or rotated) PTs with ICU duty but have not yet handled any ICU patient; and
  2. licensed PTs from JP, PH, and TW but are based and/or are working abroad.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included physical therapists who are based in Japan, Philippines, and Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Sex | November 6, 2021 to February 18, 2022
  Asked in the form of MCQ
Highest educational attainment | November 6 2021, to February 18, 2022
  PhD, Master, diploma
Work experience | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (by age range)
Hospital affiliation | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (with sub-classification: level, ownership, teaching affiliation)
ICU work experience | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (in range)
Type of ICU | November 6 2021, to February 18, 2022
  Multiple answer question
Hiring department | November 6 2021, to February 18, 2022
  Asked in the form of MCQ
Status of ICU posting | November 6 2021, to February 18, 2022
  Asked in the form of MCQ
Duration of ICU posting | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (by time range)
ICU stay per day | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (by time range)
Engagement in on-call ICU PT service | November 6 2021, to February 18, 2022
  Asked in the form of a dichotomous question
ICU PTs in the hospital | November 6 2021, to February 18, 2022
  Asked via short answer question
Source of ICU patient referral | November 6 2021, to February 18, 2022
  Asked in the form of MCQ
Number of ICU patients per day | November 6 2021, to February 18, 2022
  Asked in the form of MCQ (by range)
PT-patient ratio | November 6 2021, to February 18, 2022
  Asked in the form of MCQ
Participation in ICU-related PT trainin | November 6 2021, to February 18, 2022
  Asked in the form of dichotomus, MCQ, and multiple answer question
Most common PT techniques implemented in the ICU | November 6 2021, to February 18, 2022
  Multiple answer question
Challenges encountered in the delivery of PT services in the ICU | November 6 2021, to February 18, 2022
  Multiple answer question

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jung Cheng, PhD in BMS, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taichung, Taiwan

REFERENCES:
- [Background] Sigera PC, Tunpattu TM, Jayashantha TP, De Silva AP, Athapattu PL, Dondorp A, Haniffa R. National Profile of Physical Therapists in Critical Care Units of Sri Lanka: Lower Middle-Income Country. Phys Ther. 2016 Jul;96(7):933-9. doi: 10.2522/ptj.20150363. Epub 2016 Feb 18. PMID 26893503